CLINICAL TRIAL: NCT07085286
Title: Prognostic Value of Continuous Intra-abdominal Pressure (CIAP) and Continuous Abdominal Perfusion Pressure (CAPP) Monitoring for Acute Kidney Injury (AKI) Prediuction in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery
Brief Title: Perfusion Related Evaluation of Systemic and Renal Vulnerability to Events in CABG
Acronym: PRESERVE-CABG
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Lublin (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Manu Malbrain, Professor Critical Care Research, First Department of Anaesthesiology and Intensive Therapy, Medical University of Lublin
Other Study IDs: MUL_PRESERVE-CABG_001
Record Dates: First submitted 2025-07-06; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: AKI - Acute Kidney Injury; CABG
Keywords: abdominal pressure; IAP; abdominal perfusion pressure; mean perfusion pressure; renal perfusion pressure; prediction; AKI
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with postoperative AKI: According to KDIGO criteria
  Interventions: Device: Continous IAP measurement

INTERVENTIONS:
Device: Continous IAP measurement — Continuous IAP measurement via existing Foley bladder catheter - allowing continuous APP, MPP and RPP calculation

SUMMARY:
The goal of this observational study is to learn whether high abdominal pressure or low blood flow pressure to the kidneys is linked to kidney injury after heart surgery. The main questions it aims to answer are:

Does high abdominal pressure increase the risk of kidney injury after cardiac surgery?

Can low blood flow pressure to the kidneys help predict who may develop kidney problems?

Participants in this study are adults undergoing heart surgery, such as coronary artery bypass grafting (CABG) or valve surgery. Researchers will measure abdominal pressure and blood pressure continuously before and after surgery using medical devices that are already part of routine care. This study does not involve any changes to standard treatment.

Participants will:

Have their abdominal and blood pressures continuously monitored using existing devices

Have blood and urine tests to check kidney function

Be followed during their hospital stay and up to 30 days after surgery to assess outcomes like length of stay, readmission, and survival

This study takes place at two hospitals-one in Poland and one in the United States. Researchers hope the findings will help identify early warning signs of kidney injury and improve monitoring practices after heart surgery.

DETAILED DESCRIPTION:
This is a prospective, observational pilot study designed to investigate the relationship between elevated intra-abdominal pressure (IAP), impaired perfusion pressures, and the development of acute kidney injury (AKI) in adult patients undergoing cardiac surgery. The study will focus on whether continuous intra-abdominal pressure (CIAP) monitoring can provide early warning signs for AKI and other postoperative complications.

Intra-abdominal pressure (IAP) refers to the steady-state pressure within the abdominal cavity. In healthy individuals, IAP typically ranges between 5 and 7 millimeters of mercury (mmHg), while values may rise to around 10 mmHg in critically ill patients. Sustained IAP values at or above 12 mmHg define intra-abdominal hypertension (IAH). More severe elevations above 20 mmHg can result in abdominal compartment syndrome (ACS), which is associated with new organ dysfunction or failure. IAH can negatively impact multiple organ systems, including the kidneys, lungs, cardiovascular system, gastrointestinal tract, liver, and brain, through both mechanical and biochemical mechanisms.

Traditional IAP monitoring methods rely on intermittent measurement via the urinary bladder using a Foley catheter and saline instillation, performed at end-expiration with the patient in the supine position. Although this method is widely accepted, it is labor-intensive, operator-dependent, and cannot provide real-time pressure trends. As a result, diagnosis and management of IAH may be delayed.

Advancements in monitoring technology now allow for continuous IAP measurement using devices such as the TraumaGuard catheter. This dual-balloon Foley catheter provides real-time data on both IAP and core body temperature. It connects to standard intensive care unit (ICU) bedside monitors and allows continuous data capture and analysis.

This study will use continuous measurements of IAP, mean arterial pressure (MAP), central venous pressure (CVP), and mean alveolar pressure (Palv) to calculate key perfusion pressures:

Abdominal perfusion pressure (APP) = MAP - IAP

Mean perfusion pressure (MPP) = MAP - CVP

Renal perfusion pressure (RPP):

* In patients not receiving mechanical ventilation: RPP = MAP - IAP - CVP
* In mechanically ventilated patients: RPP = MAP - IAP - CVP - Palv

Continuous monitoring will also allow for the calculation of area under the curve (AUC) and time above threshold (TAT), providing a dynamic view of the pressure-time burden and potentially offering earlier insight into evolving complications. These data will be analyzed to assess whether sustained periods of low APP, MPP, or RPP are associated with higher rates of AKI and other adverse outcomes.

Cardiac surgery patients are considered at high risk for IAH due to fluid shifts, systemic inflammation, positive pressure ventilation, and reduced abdominal wall compliance. This study will capture multiple IAH risk factors, including patient demographics (e.g., obesity, body mass index, age), surgical variables (e.g., cardiopulmonary bypass duration, transfusion volume), and clinical factors (e.g., presence of sepsis, acidosis, or coagulopathy).

All participants will receive standard-of-care monitoring, including urinary catheters and arterial lines. The TraumaGuard catheter will be used only for data collection purposes and will not influence clinical management. No deviation from routine practice is required, and the study is entirely observational in nature.

The primary outcome is the incidence of acute kidney injury (AKI), diagnosed using Kidney Disease: Improving Global Outcomes (KDIGO) criteria. AKI will be identified by changes in serum creatinine levels and reductions in urine output during the first seven postoperative days. Secondary outcomes include myocardial injury, intensive care unit (ICU) and hospital length of stay, 30-day mortality, and hospital readmission.

Perfusion pressures (MAP, APP, MPP, RPP) will be analyzed to determine the duration and depth of hypotension relative to specific thresholds. All data will be collected continuously from bedside monitors and synchronized using timestamps to ensure accuracy. The TraumaGuard data will be integrated with beat-to-beat electronic medical record data (e.g., CapsuleTech or equivalent systems).

A total of 45 adult patients undergoing elective cardiac surgery (CABG or valve surgery) will be enrolled at two academic centers. This sample size is based on previous feasibility data and is expected to generate at least 12 AKI events, sufficient to explore statistical associations, estimate variance, and refine methodology for a larger follow-up study.

Descriptive statistics will be used to summarize perfusion pressures, with group comparisons between patients who develop AKI and those who do not. Receiver operating characteristic (ROC) curve analysis will be conducted to identify thresholds of IAP, APP, MPP, and RPP that predict AKI and other complications. A Kaplan-Meier survival analysis will be used to compare outcomes based on the presence of IAH and low perfusion pressures.

Due to the limited sample size, multivariable regression analysis will not be performed in this pilot phase.

This study aims to determine whether continuous intra-abdominal pressure monitoring can serve as a clinically valuable, noninvasive method for early detection of hemodynamic deterioration and AKI after cardiac surgery. The results may inform the design of larger-scale studies and help evaluate the potential role of IAP monitoring as a new vital sign in critical care.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older
* Undergoing cardiac surgery (CABG, valve surgery, combined procedures, heart transplantation, or placement of assist device)
* Expected hospital stay of at least one night
* Preoperative serum creatinine measurement available
* At least one postoperative serum creatinine measurement available

Exclusion Criteria

* Age below 18 years
* Incarcerated individuals
* No requirement for urinary catheter placement
* Presence of a do-not-resuscitate (DNR) order
* Pregnant or lactating individuals
* Fewer than 12 hours of recorded data (including intraoperative data)
* No informed consent (if a waiver is not granted)
* Pre-existing chronic kidney disease, defined as estimated glomerular filtration rate <60 mL/min/1.73 m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This two-center prospective observational study will enroll adult patients undergoing cardiac surgery (e.g., coronary artery bypass grafting, valve surgery, or assist device placement). Participants will receive a TraumaGuard urinary catheter, which functions both as a standard Foley catheter and as a device for continuous intra-abdominal pressure monitoring. Data will be collected during and after surgery. An initial cohort of 45 patients will be analyzed for feasibility and to inform the sample size for future enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury (AKI) in participants with and without intra-abdominal hypertension (IAH) | Postoperative Days 0 through 7
  To determine whether the presence of intra-abdominal hypertension (IAP ≥ 12 mmHg) is associated with a higher incidence of AKI follow.
  Measure Type: Binary outcome. Unit of Measure: % of participants with AKI. Method of Assessment: AKI will be diagnosed using the Kidney Disease: Improving Global Outcomes (KDIGO) criteria, based on changes in serum creatinine and urine output. IAH will be defined as intra-abdominal pressure (IAP) ≥ 12 mmHg, measured using continuous intra-abdominal pressure monitoring.

SECONDARY OUTCOMES:
Association between abdominal perfusion pressure (APP) and incidence of acute kidney injury (AKI) | Postoperative Days 0 through 7
  To assess whether lower abdominal perfusion pressure (APP = mean arterial pressure - intra-abdominal pressure) is associated with a higher risk of AKI.
  Measure Type: Comparative association. Unit of Measure: Odds ratio for AKI or % of participants with AKI by APP range. Method of Assessment: APP will be calculated using continuously recorded mean arterial pressure (MAP) and intra-abdominal pressure (IAP). AKI will be assessed using KDIGO criteria.
Association between mean perfusion pressure (MPP) and incidence of acute kidney injury (AKI) | Postoperative Days 0 through 7
  To assess whether lower mean perfusion pressure (MPP = mean arterial pressure - central venous pressure) is associated with a higher risk of AKI.
  Measure Type: Comparative association. Unit of Measure: Odds ratio for AKI or % of participants with AKI by MPP range. Method of Assessment: MPP will be calculated using continuously recorded mean arterial pressure (MAP) and central venous pressure (CVP). AKI will be assessed using KDIGO criteria.
Association between renal perfusion pressure (RPP) and incidence of acute kidney injury (AKI) | Postoperative Days 0 through 7
  To evaluate whether lower renal perfusion pressure (RPP) is associated with an increased risk of AKI after cardiac surgery.
  In non-ventilated patients: RPP = MAP - IAP - CVP
  In mechanically ventilated patients: RPP = MAP - IAP - CVP - mean alveolar pressure (Palv) Measure Type: Comparative association. Unit of Measure: Odds ratio for AKI or % of participants with AKI by RPP range. Method of Assessment: RPP will be calculated using continuously recorded mean arterial pressure (MAP), intra-abdominal pressure (IAP), central venous pressure (CVP), and mean alveolar pressure (Palv) where applicable. AKI is defined using KDIGO criteria.
Association between intra-abdominal hypertension (IAH) and postoperative myocardial injury | Postoperative Days 0 through 7
  To evaluate whether participants who develop intra-abdominal hypertension (IAP ≥ 12 mmHg) are more likely to experience myocardial injury after cardiac surgery.
  Measure Type: Binary outcome. Unit of Measure: % of participants with myocardial injury. Method of Assessment: Myocardial injury defined by cardiac biomarkers: troponin T ≥ 0.04 µg/L or creatine kinase-MB (CK-MB) ≥ 8.8 ng/mL, measured within 7 days of surgery.
Agreement between intra-abdominal pressure (IAP) measurements using the TraumaGuard device and standard intermittent bladder pressure measurements | Up to 48 hours post-surgery (duration of Foley catheter placement in ICU)
  To assess the agreement, accuracy, and reliability of intra-abdominal pressure (IAP) monitoring using the TraumaGuard catheter (IAPTG) compared to the gold-standard intermittent transvesical measurement technique. Agreement will be evaluated using statistical measures such as Bland-Altman plots and intraclass correlation coefficients (ICC).
  Measure Type: Comparative diagnostic performance. Unit of Measure: Intraclass correlation coefficient (ICC), mean difference (mmHg), limits of agreement (mmHg).
  Method of Assessment: Intra-abdominal pressure will be measured simultaneously using both the TraumaGuard catheter system and the intermittent bladder pressure method. Measurements will be recorded at predefined intervals with the patient in supine position. Agreement between methods will be analyzed to determine validity, reproducibility, and potential clinical interc

IPD SHARING:
Plan to Share IPD: Undecided
Needs to be defined

REFERENCES:
- [Background] Dang PT, Lopez BE, Togashi K. A Decrease in Effective Renal Perfusion Pressure Is Associated With Increased Acute Kidney Injury in Patients Undergoing Cardiac Surgery. Cureus. 2023 Sep 11;15(9):e45036. doi: 10.7759/cureus.45036. eCollection 2023 Sep. PMID 37829983
- [Background] Goeddel LA, Hernandez M, Koffman L, Murphy Z, Khanna AK, Robich M, Whitman G, Zhou X, Bandeen-Roche K, Muschelli J 3rd, Parikh CR, Lima JAC, Crainiceanu CM, Brown C 4th, Faraday N. Fine-Mapping the Association of Acute Kidney Injury With Mean Arterial and Central Venous Pressures During Coronary Artery Bypass Surgery. Anesth Analg. 2025 Jun 1;140(6):1439-1449. doi: 10.1213/ANE.0000000000007500. Epub 2025 Apr 17. PMID 40244889
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Kopitko C, Medve L, Gondos T. The value of combined hemodynamic, respiratory and intra-abdominal pressure monitoring in predicting acute kidney injury after major intraabdominal surgeries. Ren Fail. 2019 Nov;41(1):150-158. doi: 10.1080/0886022X.2019.1587467. PMID 30909772
- [Background] Cheatham ML, White MW, Sagraves SG, Johnson JL, Block EF. Abdominal perfusion pressure: a superior parameter in the assessment of intra-abdominal hypertension. J Trauma. 2000 Oct;49(4):621-6; discussion 626-7. doi: 10.1097/00005373-200010000-00008. PMID 11038078
- [Background] Panwar R, Tarvade S, Lanyon N, Saxena M, Bush D, Hardie M, Attia J, Bellomo R, Van Haren F; REACT Shock Study Investigators and Research Coordinators. Relative Hypotension and Adverse Kidney-related Outcomes among Critically Ill Patients with Shock. A Multicenter, Prospective Cohort Study. Am J Respir Crit Care Med. 2020 Nov 15;202(10):1407-1418. doi: 10.1164/rccm.201912-2316OC. PMID 32614244
- [Background] Schneider AG, Goodwin MD, Bellomo R. Measurement of kidney perfusion in critically ill patients. Crit Care. 2013 Mar 19;17(2):220. doi: 10.1186/cc12529. No abstract available. PMID 23514525
- [Background] Mullens W, Abrahams Z, Francis GS, Sokos G, Taylor DO, Starling RC, Young JB, Tang WHW. Importance of venous congestion for worsening of renal function in advanced decompensated heart failure. J Am Coll Cardiol. 2009 Feb 17;53(7):589-596. doi: 10.1016/j.jacc.2008.05.068. PMID 19215833
- [Background] Loutzenhiser R, Griffin K, Williamson G, Bidani A. Renal autoregulation: new perspectives regarding the protective and regulatory roles of the underlying mechanisms. Am J Physiol Regul Integr Comp Physiol. 2006 May;290(5):R1153-67. doi: 10.1152/ajpregu.00402.2005. PMID 16603656
- [Background] Malbrain MLNG, Tantakoun K, Zara AT, Ferko NC, Kelly T, Dabrowski W. Urine output is an early and strong predictor of acute kidney injury and associated mortality: a systematic literature review of 50 clinical studies. Ann Intensive Care. 2024 Jul 9;14(1):110. doi: 10.1186/s13613-024-01342-x. PMID 38980557
- [Background] Chawla LS, Bellomo R, Bihorac A, Goldstein SL, Siew ED, Bagshaw SM, Bittleman D, Cruz D, Endre Z, Fitzgerald RL, Forni L, Kane-Gill SL, Hoste E, Koyner J, Liu KD, Macedo E, Mehta R, Murray P, Nadim M, Ostermann M, Palevsky PM, Pannu N, Rosner M, Wald R, Zarbock A, Ronco C, Kellum JA; Acute Disease Quality Initiative Workgroup 16.. Acute kidney disease and renal recovery: consensus report of the Acute Disease Quality Initiative (ADQI) 16 Workgroup. Nat Rev Nephrol. 2017 Apr;13(4):241-257. doi: 10.1038/nrneph.2017.2. Epub 2017 Feb 27. PMID 28239173
- [Background] O'Neal JB, Shaw AD, Billings FT 4th. Acute kidney injury following cardiac surgery: current understanding and future directions. Crit Care. 2016 Jul 4;20(1):187. doi: 10.1186/s13054-016-1352-z. PMID 27373799
- [Background] Han SS, Shin N, Baek SH, Ahn SY, Kim DK, Kim S, Chin HJ, Chae DW, Na KY. Effects of acute kidney injury and chronic kidney disease on long-term mortality after coronary artery bypass grafting. Am Heart J. 2015 Mar;169(3):419-25. doi: 10.1016/j.ahj.2014.12.019. Epub 2015 Jan 6. PMID 25728733
- [Background] Drosos G, Ampatzidou F, Sarafidis P, Karaiskos T, Madesis A, Boutou AK. Serum Creatinine and Chronic Kidney Disease-Epidemiology Estimated Glomerular Filtration Rate: Independent Predictors of Renal Replacement Therapy following Cardiac Surgery. Am J Nephrol. 2018;48(2):108-117. doi: 10.1159/000492182. Epub 2018 Aug 15. PMID 30110680
- [Background] Chew STH, Hwang NC. Acute Kidney Injury After Cardiac Surgery: A Narrative Review of the Literature. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):1122-1138. doi: 10.1053/j.jvca.2018.08.003. Epub 2018 Aug 7. PMID 30228051
- [Background] Machado MN, Nakazone MA, Maia LN. Prognostic value of acute kidney injury after cardiac surgery according to kidney disease: improving global outcomes definition and staging (KDIGO) criteria. PLoS One. 2014 May 14;9(5):e98028. doi: 10.1371/journal.pone.0098028. eCollection 2014. PMID 24826910
- [Background] Bastin AJ, Ostermann M, Slack AJ, Diller GP, Finney SJ, Evans TW. Acute kidney injury after cardiac surgery according to Risk/Injury/Failure/Loss/End-stage, Acute Kidney Injury Network, and Kidney Disease: Improving Global Outcomes classifications. J Crit Care. 2013 Aug;28(4):389-96. doi: 10.1016/j.jcrc.2012.12.008. Epub 2013 Jun 3. PMID 23743540
- [Background] Khanna AK, Rola P, Malbrain MLNG. Biomarkers for intra-abdominal pressure: another tool in the toolbox? Eur Heart J Acute Cardiovasc Care. 2022 Jun 22;11(6):461-463. doi: 10.1093/ehjacc/zuac073. No abstract available. PMID 35695764
- [Background] Tayebi S, McKinney T, McKinney C, Delvadia D, Levine MA, Spofford ES Jr, Malbrain L, Stiens J, Dabrowski W, Malbrain MLNG. Evaluation of the TraumaGuard Balloon-in-Balloon Catheter Design for Intra-Abdominal Pressure Monitoring: Insights from Pig and Human Cadaver Studies. Sensors (Basel). 2023 Oct 29;23(21):8806. doi: 10.3390/s23218806. PMID 37960507
- [Background] Tayebi S, Wise R, Pourkazemi A, Stiens J, Malbrain MLNG. Pre-Clinical Validation of A Novel Continuous Intra-Abdominal Pressure Measurement Equipment (SERENNO). Life (Basel). 2022 Jul 30;12(8):1161. doi: 10.3390/life12081161. PMID 36013340
- [Background] Malbrain MLNG, De Keulenaer BL, Khanna AK. Continuous intra-abdominal pressure: is it ready for prime time? Intensive Care Med. 2022 Oct;48(10):1501-1504. doi: 10.1007/s00134-022-06780-4. Epub 2022 Aug 4. No abstract available. PMID 35925322
- [Background] De Potter TJ, Dits H, Malbrain ML. Intra- and interobserver variability during in vitro validation of two novel methods for intra-abdominal pressure monitoring. Intensive Care Med. 2005 May;31(5):747-51. doi: 10.1007/s00134-005-2597-1. Epub 2005 Apr 5. PMID 15809871
- [Background] Malbrain ML, De laet I, Viaene D, Schoonheydt K, Dits H. In vitro validation of a novel method for continuous intra-abdominal pressure monitoring. Intensive Care Med. 2008 Apr;34(4):740-5. doi: 10.1007/s00134-007-0952-0. Epub 2007 Dec 13. PMID 18075730
- [Background] Malbrain ML. Different techniques to measure intra-abdominal pressure (IAP): time for a critical re-appraisal. Intensive Care Med. 2004 Mar;30(3):357-71. doi: 10.1007/s00134-003-2107-2. Epub 2004 Jan 17. PMID 14730376
- [Background] Czajkowski M, Dabrowski W. Changes in intra-abdominal pressure during CABG with normovolemic hemodilution. Med Sci Monit. 2006 Nov;12(11):CR487-92. PMID 17072275
- [Background] Dabrowski W, Rola P, Malbrain MLNG. Intra-abdominal pressure monitoring in cardiac surgery: is this the canary in the coalmine for kidney injury? J Clin Monit Comput. 2023 Apr;37(2):351-358. doi: 10.1007/s10877-022-00933-y. Epub 2022 Dec 22. No abstract available. PMID 36550345
- [Background] Moll V, Khanna AK, Kurz A, Huang J, Smit M, Swaminathan M, Minear S, Parr KG, Prabhakar A, Zhao M, Malbrain MLNG. Optimization of kidney function in cardiac surgery patients with intra-abdominal hypertension: expert opinion. Perioper Med (Lond). 2024 Jul 12;13(1):72. doi: 10.1186/s13741-024-00416-5. PMID 38997752
- [Background] Khanna AK, Minear S, Kurz A, Moll V, Stanton K, Essakalli L, Prabhakar A; Predict AKI Group. Intra-abdominal hypertension in cardiac surgery patients: a multicenter observational sub-study of the Accuryn registry. J Clin Monit Comput. 2023 Feb;37(1):189-199. doi: 10.1007/s10877-022-00878-2. Epub 2022 Jun 13. PMID 35695943
- [Background] Malbrain ML. Abdominal pressure in the critically ill: measurement and clinical relevance. Intensive Care Med. 1999 Dec;25(12):1453-8. doi: 10.1007/s001340051098. No abstract available. PMID 10702030
- [Background] Reintam Blaser A, Regli A, De Keulenaer B, Kimball EJ, Starkopf L, Davis WA, Greiffenstein P, Starkopf J; Incidence, Risk Factors, and Outcomes of Intra-Abdominal (IROI) Study Investigators. Incidence, Risk Factors, and Outcomes of Intra-Abdominal Hypertension in Critically Ill Patients-A Prospective Multicenter Study (IROI Study). Crit Care Med. 2019 Apr;47(4):535-542. doi: 10.1097/CCM.0000000000003623. PMID 30608280
- [Background] Wise R, Jacobs J, Pilate S, Jacobs A, Peeters Y, Vandervelden S, Van Regenmortel N, De Laet I, Schoonheydt K, Dits H, Malbrain ML. Incidence and prognosis of intra-abdominal hypertension and abdominal compartment syndrome in severely burned patients: Pilot study and review of the literature. Anaesthesiol Intensive Ther. 2016;48(2):95-109. doi: 10.5603/AIT.a2015.0083. Epub 2015 Nov 20. PMID 26588479
- [Background] Malbrain ML, Chiumello D, Pelosi P, Bihari D, Innes R, Ranieri VM, Del Turco M, Wilmer A, Brienza N, Malcangi V, Cohen J, Japiassu A, De Keulenaer BL, Daelemans R, Jacquet L, Laterre PF, Frank G, de Souza P, Cesana B, Gattinoni L. Incidence and prognosis of intraabdominal hypertension in a mixed population of critically ill patients: a multiple-center epidemiological study. Crit Care Med. 2005 Feb;33(2):315-22. doi: 10.1097/01.ccm.0000153408.09806.1b. PMID 15699833
- [Background] Reintam A, Parm P, Kitus R, Starkopf J, Kern H. Gastrointestinal failure score in critically ill patients: a prospective observational study. Crit Care. 2008;12(4):R90. doi: 10.1186/cc6958. Epub 2008 Jul 14. PMID 18625051
- [Background] Bongard F, Pianim N, Dubecz S, Klein SR. Adverse consequences of increased intra-abdominal pressure on bowel tissue oxygen. J Trauma. 1995 Sep;39(3):519-24; discussion 524-5. doi: 10.1097/00005373-199509000-00020. PMID 7473918
- [Background] Diebel LN, Dulchavsky SA, Wilson RF. Effect of increased intra-abdominal pressure on mesenteric arterial and intestinal mucosal blood flow. J Trauma. 1992 Jul;33(1):45-8; discussion 48-9. doi: 10.1097/00005373-199207000-00010. PMID 1635105
- [Background] Diebel LN, Dulchavsky SA, Brown WJ. Splanchnic ischemia and bacterial translocation in the abdominal compartment syndrome. J Trauma. 1997 Nov;43(5):852-5. doi: 10.1097/00005373-199711000-00019. PMID 9390500
- [Background] Malbrain ML, Viaene D, Kortgen A, De Laet I, Dits H, Van Regenmortel N, Schoonheydt K, Bauer M. Relationship between intra-abdominal pressure and indocyanine green plasma disappearance rate: hepatic perfusion may be impaired in critically ill patients with intra-abdominal hypertension. Ann Intensive Care. 2012 Dec 20;2 Suppl 1(Suppl 1):S19. doi: 10.1186/2110-5820-2-S1-S19. Epub 2012 Dec 20. PMID 23282242
- [Background] Cresswell AB, Wendon JA. Hepatic function and non-invasive hepatosplanchnic monitoring in patients with abdominal hypertension. Acta Clin Belg. 2007;62 Suppl 1:113-8. doi: 10.1179/acb.2007.62.s1.014. PMID 24881707
- [Background] De Waele JJ, De Laet I, Kirkpatrick AW, Hoste E. Intra-abdominal Hypertension and Abdominal Compartment Syndrome. Am J Kidney Dis. 2011 Jan;57(1):159-69. doi: 10.1053/j.ajkd.2010.08.034. PMID 21184922
- [Background] De Laet I, Malbrain ML, Jadoul JL, Rogiers P, Sugrue M. Renal implications of increased intra-abdominal pressure: are the kidneys the canary for abdominal hypertension? Acta Clin Belg. 2007;62 Suppl 1:119-30. doi: 10.1179/acb.2007.62.s1.015. PMID 24881708
- [Background] Regli A, Pelosi P, Malbrain MLNG. Ventilation in patients with intra-abdominal hypertension: what every critical care physician needs to know. Ann Intensive Care. 2019 Apr 25;9(1):52. doi: 10.1186/s13613-019-0522-y. PMID 31025221
- [Background] Pelosi P, Quintel M, Malbrain ML. Effect of intra-abdominal pressure on respiratory mechanics. Acta Clin Belg. 2007;62 Suppl 1:78-88. PMID 17469705
- [Background] De Laet I, Citerio G, Malbrain ML. The influence of intra-abdominal hypertension on the central nervous system: current insights and clinical recommendations, is it all in the head? Acta Clin Belg. 2007;62 Suppl 1:89-97. doi: 10.1179/acb.2007.62.s1.012. PMID 24881705
- [Background] Malbrain ML, De Waele JJ, De Keulenaer BL. What every ICU clinician needs to know about the cardiovascular effects caused by abdominal hypertension. Anaesthesiol Intensive Ther. 2015;47(4):388-99. doi: 10.5603/AIT.a2015.0028. Epub 2015 May 14. PMID 25973663
- [Background] Cheatham ML, Malbrain ML. Cardiovascular implications of abdominal compartment syndrome. Acta Clin Belg. 2007;62 Suppl 1:98-112. PMID 17469707
- [Background] Malbrain ML, Chiumello D, Cesana BM, Reintam Blaser A, Starkopf J, Sugrue M, Pelosi P, Severgnini P, Hernandez G, Brienza N, Kirkpatrick AW, Schachtrupp A, Kempchen J, Estenssoro E, Vidal MG, De Laet I, De Keulenaer BL. A Systematic Review And Individual Patient Data Meta-Analysis On Intraabdominal Hypertension In Critically Ill Patients: The Wake-Up Project World Initiative on Abdominal Hypertension Epidemiology, a Unifying Project (WAKE-Up!). Minerva Anestesiol. 2013 Dec 12. Online ahead of print. PMID 24336093
- [Background] Malbrain ML. Is it wise not to think about intraabdominal hypertension in the ICU? Curr Opin Crit Care. 2004 Apr;10(2):132-45. doi: 10.1097/00075198-200404000-00010. PMID 15075724
- [Background] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399